## Activating and Connecting Teens (ACT) Study NCT03438656 03/01/2021

## **ACT Study Protocol and Statistical Analysis Plan**

Childhood maltreatment is common<sup>1,2</sup> and has been linked to a multitude of negative outcomes, including psychiatric and functional impairments that persist across the lifespan.<sup>2–4</sup> Exposure to physical, sexual, or emotional abuse or neglect is associated with markedly elevated risk for depression<sup>5</sup> with epidemiological studies indicating that these forms of childhood maltreatment (CM) account for as much as 30% of depression onsets in the population<sup>2,6</sup> and predict a more chronic and severe course of depression.<sup>7</sup> Currently cognitive behavioral therapy and antidepressant medication is recommended as best practice for treatment of depression.<sup>8</sup> However, depressed individuals who have experienced CM show poor treatment response and high risk for relapse across interventions,<sup>7,9–11</sup> and **alternative treatments have not been investigated**.

A history of CM exposure may increase risk for depression via altered neurodevelopment of the **positive valence system** (i.e., reward processing). Given the reward processing deficits observed among depressed youth with a history of CM exposure, depression outcomes may be improved by investigating interventions that specifically target disruptions in reward circuitry and behaviors.

Behavioral Activation (BA) is an evidence-based treatment for adult and adolescent depression <sup>13–15</sup> that uses an individualized approach to identify and foster behaviors within an adolescent's context that increase rewarding experiences and decrease avoidant behaviors that contribute to depression symptom severity and maintenance. This is the first study to investigate BA as an alternative, target-focused approach to treat depression among adolescents with a history of CM exposure.

This proposal will examine whether BA intervention reduces depression and anhedonia in a sample of depressed adolescents, aged 13-18, with variable histories of CM exposure (**BA Group**). A total of 30 depressed adolescents will be recruited to undergo a 12-week course of BA. All participants will undergo clinical assessment to measure depression symptoms and anhedonia at baseline (Week 0) and post- (Week 12) treatment.

| Participant Table | Inclusion Criteria | Exclusion Criteria |
|---|---|---|
| | 1) Age 13-18; 2) major or minor | 1) IQ<80; 2) non-English speaking; 3) current |
| BA Group n=30 | depression (PHQ ≥10). | PTSD; 4) developmental, neurological, psychosis, |
| | | bipolar, or substance disorder; 5) No legal |
| | | guardian; 6) current psychiatric medication; 7) |
| | | suicidality requiring higher level of care. |

## **Study Aims:**

<u>Aim 1:</u> Determine baseline and post-BA treatment depression and anhedonia symptoms among depressed adolescents with variable histories of CM.

**Exploratory Aim:** Evaluate whether changes in self-reported anhedonia or other indicators of reward processing as measured by daily ecological momentary assessment and self-report are differentially associated with reductions in depression following BA in youth with versus without CM exposure.

**Data Analyses:** Across all analyses: *primary outcomes* will be measured as 1) depression and anhedonia symptoms. **Aim 1. Determine baseline and post-BA treatment depression and anhedonia symptoms among depressed adolescents with variable histories of CM.** Means and standard deviations in depression (PHQ-9) and anhedonia symptoms (BADS) will be measured at baseline and post-treatment follow-up.

**Exploratory aim**. Evaluate whether changes in self-reported anhedonia or other indicators of reward processing are differentially associated with reductions in depression following BA in youth with versus without CM exposure. Participants completed morning, afternoon, and evening EMA surveys twice a week over 14 weeks (n= 84 timepoints). Measures assessed depression symptoms, CM exposure, and reward processing/responsiveness across BA treatment. Using the *lavaan* package in R<sup>8</sup>, we plan to conduct Latent Growth Modeling (LGM) to test the associations between changes in reward processing and depression symptoms with CM as a fixed moderator. Covariates will include age, sex, and socioeconomic status.

## References

- 1. Green JG, McLaughlin KA, Berglund PA, et al. Childhood adversities and adult psychiatric disorders in the national comorbidity survey replication I: associations with first onset of DSM-IV disorders. *Arch Gen Psychiatry*. 2010;67(2):113-123.
- McLaughlin KA, Green JG, Gruber MJ, Sampson NA, Zaslavsky AM, Kessler RC. Childhood adversities and first onset of psychiatric disorders in a national sample of US adolescents. Arch Gen Psychiatry. 2012;69(11):1151-1160.
- 3. McLaughlin KA, Green JG, Gruber MJ, Sampson NA, Zaslavsky AM, Kessler RC. Childhood adversities and adult psychiatric disorders in the national comorbidity survey replication II: associations with persistence of DSM-IV disorders. *Arch Gen Psychiatry*. 2010;67(2):124-132.
- 4. McLaughlin KA, Green JG, Gruber MJ, Sampson NA, Zaslavsky AM, Kessler RC. Childhood adversities and adult psychopathology in the National Comorbidity Survey Replication (NCS-R) III: associations with functional impairment related to DSM-IV disorders. *Psychol Med*. 2010;40(05):847-859.
- 5. Kessler RC. The effects of stressful life events on depression. *Annu Rev Psychol.* 1997;48:191-214. doi:10.1146/annurev.psych.48.1.191
- 6. Affif TO, Boman J, Fleisher W, Sareen J. The relationship between child abuse, parental divorce, and lifetime mental disorders and suicidality in a nationally representative adult sample. *Child Abuse Negl.* 2009;33(3):139-147.
- 7. Nanni V, Uher R, Danese A. Childhood Maltreatment Predicts Unfavorable Course of Illness and Treatment Outcome in Depression: A Meta-Analysis. *Am J Psychiatry*. 2012;169(2):141-151. doi:10.1176/appi.ajp.2011.11020335
- 8. Birmaher B, Brent D. Practice Parameter for the Assessment and Treatment of Children and Adolescents With Depressive Disorders. *J Am Acad Child Adolesc Psychiatry*. 2007;46(11):1503-1526. doi:10.1097/chi.0b013e318145ae1c
- 9. Lewis CC, Simons AD, Nguyen LJ, et al. Impact of childhood trauma on treatment outcome in the Treatment for Adolescents with Depression Study (TADS). *J Am Acad Child Adolesc Psychiatry*. 2010;49(2):132-140.
- Brent DA, Emslie GJ, Clarke GN, et al. Predictors of spontaneous and systematically assessed suicidal adverse events in the treatment of SSRI-resistant depression in adolescents (TORDIA) study. Am J Psychiatry. 2009;166(4):418-426.
- 11. Shamseddeen W, Asarnow JR, Clarke G, et al. Impact of physical and sexual abuse on treatment response in the Treatment of Resistant Depression in Adolescent Study (TORDIA). *J Am Acad Child Adolesc Psychiatry*. 2011;50(3):293-301.
- 12. Dillon DG, Holmes AJ, Birk JL, Brooks N, Lyons-Ruth K, Pizzagalli DA. Childhood adversity is associated with left basal ganglia dysfunction during reward anticipation in adulthood. *Biol Psychiatry*. 2009;66(3):206-213.
- 13. Richardson L, McCauley E, Katon W. Collaborative care for adolescent depression: a pilot study. *Gen Hosp Psychiatry*. 2009;31(1):36-45. doi:10.1016/j.genhosppsych.2008.09.019
- 14. Cuijpers P, van Straten A, Warmerdam L. Behavioral activation treatments of depression: A meta-analysis. *Clin Psychol Rev.* 2007;27(3):318-326. doi:10.1016/j.cpr.2006.11.001
- 15. McCauley E, Gudmundsen G, Schloredt K, et al. The Adolescent Behavioral Activation Program: Adapting Behavioral Activation as a Treatment for Depression in Adolescence. *J Clin Child Adolesc Psychol*. Published online 2015. doi:10.1080/15374416.2014.979933